CLINICAL TRIAL: NCT05731466
Title: Exercise Measurement of Right Ventricular-arterial Coupling to Predict Hemodynamic Worsening in Heart Failure and Preserved Ejection Fraction
Brief Title: Exercise Right Ventricular Coupling in HFpEF
Acronym: ENDURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, dr. Guido Claessen, Clinical Professor - Principal Investigator (MD. PhD), Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDURE
Record Dates: First submitted 2022-12-21; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Pulmonary Hypertension
Keywords: CardioMems; Exercise cardiovascular magnetic resonance; Heart Failure with Preserved Ejection Fraction; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CardioMems (Clinical Indication) (Other): Single Arm, CardioMems implantation on clinical indication. No control group. Every participant is his/her own control (longitudinal follow-up)
  Interventions: Device: CardioMems HF System

INTERVENTIONS:
Device: CardioMems HF System — 1. Implantation CardioMems device.
  2. Evaluation of right ventricular-arterial coupling during exercise using a hybrid technique of real-time CMR-derived volume measures and CardioMems-derived pulmonary artery pressure measurements.
  Other Names: CMR

SUMMARY:
The investigators aim to evaluate the feasibility and prognostic value of right ventricular-arterial coupling (RVAC) during exercise in patients with HFpEF-PH using a hybrid technique of real-time CMRderived volume measures and CardioMEMS-derived pulmonary artery pressure measurements.

The investigators will determine:

1. Whether exercise RV-arterial coupling at baseline (assessed using hybrid CMRCardioMEMS) predicts development or worsening of exercise RV-arterial uncoupling during follow-up in HFpEF-PH patients.
2. If HFpEF-PH patients developing RV dysfunction have a particular PAP pattern as assessed remotely using the CardioMEMS system. The investigators will determine differential characteristics in CardioMEMS pressure patterns in those developing RV dysfunction versus those who do not develop RV dysfunction, both at rest and during exercise. Hence, HFpEF-PH patients developing RV dysfunction may harbor a plateau of pulmonary artery pressures (as a reflection of RV-arterial uncoupling) despite clinical worsening.
3. Whether extraction of raw pressure data obtained by the CardioMEMS system is feasible and enables post-processing using machine learning methods (artificial intelligence) for deep phenotyping of patients (in addition to clinical evaluation of pressure waveforms).

The investigators aim to evaluate the effect of SGLT-2 inhibitors on RV-arterial coupling in patients with HFpEF-PH. In case a patient is not using an SGLT-2 inhibitor, the investigators will prescribe this after baseline testing, since SGLT-2 inhibitors are clinically indicated in these patients.

DETAILED DESCRIPTION:
In this prospective, two-center study, the investigators will recruit 30 HFpEF-PH patients in whom a CardioMEMS device will be implanted because of clinical indication. Potential study candidates will be enrolled in the outpatient clinic or during hospitalization.

Subjects who sign the informed consent form and meet the eligibility criteria at the baseline visit will be eligible for the trial. Subjects will undergo the study-related procedures, including clinical laboratory measurements and body mass index (BMI) calculation.

Eligible subjects will be scheduled for the Implant procedure (PA sensor implant in conjunction with a RHC procedure).

Subjects must also have an appropriately sized (≥7mm diameter) pulmonary artery branch identified by a selective pulmonary angiogram prior to Sensor implant. Subjects who do not meet this inclusion criteria will be documented as consented not implanted.

After implantation of the CardioMEMS device, the patient will be asked to perform cardiopulmonary exercise testing (CPET) with continuous expiratory gas monitoring on an upright cycle ergometer (ER900 and Alpha, Jaeger, Germany), using a continuous ramp protocol until exhaustion.

During the next visit, exercise RVAC will be assessed using a hybrid approach of exercise CMR and PAP measurement using the CardioMEMS system (Figure 1). Firstly, subjects will perform supine bicycle exercise within the CMR bore using a cycle-ergometer with adjustable electronic resistance (Lode, Groningen, The Netherlands). Exercise workloads for the exercise CMR protocol will be determined as 25%, 50% and 66% of peak power (Pmax) achieved during previous CPET, as the investigators previously demonstrated that supine exercise at 66% of peak power closely corresponds to maximal sustainable exercise intensity in an upright position. After the exercise test in the CMR bore, a second exercise test will be repeated on a supine bicycle ergometer. The CardioMEMS transmit-receive coil will be put under the back of the supine patient. After waiting one minute for the patient to stabilize, the CardioMEMS measurement will be initiated at rest and subsequently at the same workloads as during the exercise CMR protocol. This second exercise test will be combined with a exercise echocardiography.

CMR imaging will be performed on a Philips 1.5T CMR (Philips Medical Systems, Best, The Netherlands). RV-arterial coupling will be evaluated using a combined approach of CardioMEMS-derived pulmonary artery pressure data and CMR-derived volume data, thereby enabling the calculation of RV end-systolic pressure volume relationships. In addition, RVEF will be assessed as surrogate measure of RV-arterial coupling.

Prior to hospital discharge, subjects will be trained on the home monitoring system and instructed to take pulmonary artery pressure measurements daily at approximately the same time each day in the morning or as directed by their physician. Subjects will be supplied with a patient implant identification card, a Patient System Manual, and a Helpline phone number.

After discharge, the subject will take PA pressure measurements at home, as directed by the investigator, utilizing the CardioMEMS HF System. These measurements will be transmitted via modem to a secure data base. Patient compliance will be monitored by the Investigator.

Follow-up study visits will be scheduled at Month 1, Month 6, and every 6 months thereafter for 2 years (± 14 days visit window). Follow-up visits will include a physical exam, evaluation of NYHA Class, heart failure medications review, quality of life assessment, and assessment of any hospitalizations (including HF hospitalizations), that may have occurred between visits. In addition, all contacts between site staff and study subjects post implant will be recorded on a log to capture frequency, purpose and outcome of each contact.

The hybrid exercise CMR-CardioMEMS-derived assessment of exercise RVAC will be repeated at Month 6 and after 1 year following the same exercise protocol as detailed above.

All subjects included in this trial meet the criteria to start a SGLT-2 inhibitor on clinical indication following the latest evidence. Those who currently lack a SGLT-2 inhibitor, this medication will be initiated after the run-in period and the baseline testing (6 weeks after implantation of de CardioMems device).

Biochemistry will involve traditional parameters, such as hemoglobin, hematocrit, ionogram, renal function, NTproBNP, hs-troponin hs-CRP, ferritin, transferrin and iron level. In addition, at each time point, samples (serum and whole blood) will be stored for future analyses at Biobank UZ Leuven.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from subject
2. > 18 years of age
3. Diagnosis of NYHA Class III Heart Failure with preserved ejection fraction defined as LVEF≥45%
4. At least 1 heart failure related hospitalization or urgent outpatient visit within 12 months of baseline visit
5. Presence of pulmonary hypertension defined as mPAP>25 mmHg at rest or mPAP/CO slope >3 mmHg/L/min during exercise during right heart catheterization or tricuspid regurgitation velocity of > 2.8 m/s assessed by transthoracic echocardiography (data must be taken within the last 6 months prior to implantation)
6. Subjects with a BMI ≤ 35. Subjects with BMI >35 will require their chest circumference to be measured at the axillary level, if > 65 inches the patient will not be eligible for the study.
7. Subjects with pulmonary artery branch diameter ≥ 7mm - (implant target artery - assessed during the RHC)
8. Subjects willing and able to comply with the follow-up requirements of the study
9. All participants need to be able to perform at least 40 watts on an upright bicycle stress test.

Exclusion Criteria:

1. Subjects with an active infection
2. Subjects with history of recurrent (> 1) pulmonary embolism or deep vein thrombosis
3. Subjects who, in the Investigator's opinion, are unable to tolerate a right heart catheterization
4. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, open heart surgery, stroke, etc.) within 2 months of Baseline Visit
5. Subjects with Cardiac Resynchronization Device (CRT) , pacemaker or Implantable Cardioverter Defibrillator (ICD)
6. Subjects with a Glomerular Filtration Rate (GFR) < 25 ml/min (obtained within 2 weeks of the baseline visit) who are non-responsive to diuretic therapy or who are on chronic renal dialysis
7. Subjects with congenital heart disease or mechanical heart valve(s)
8. Subjects likely to undergo heart transplantation or VAD within 6 months of baseline visit
9. Subjects with known coagulation disorders
10. Subjects with a hypersensitivity or allergy to aspirin, and/or clopidogrel (not applicable for subjects taking anti-coagulation therapy or other approved anti-platelets therapy).
11. Subjects with history of coronary artery bypass surgery (CABG)
12. Subjects with severe valvular disease (4/4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-10-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Right ventricular-arterial coupling (RVAC) | 12 months
  Whether baseline exercise RV-arterial coupling, determined by exercise CMR-CardioMems, can predict the development of progressive RV dysfunction after one year

SECONDARY OUTCOMES:
VO2max (mL/kg/min) | 12 months
  Evaluation whether exercise RV-arterial uncoupling is associated with clinical worsening by a relative VO2max ≥6% change (i.e. change of VO2max (ml/kg/min) from baseline to follow-up)
Right heart failure hospitalisation | 12 months
  Number of participants with the combined secondary endpoint of (1) hospitalization for right heart failure requiring intravenous diuretics or (2) death from any cause
SGLT-2 | 12 months
  Whether initiation of a SGLT-2 inhibitor, after baseline evaluation, has a positive effect on exercise RV-arterial coupling at one year of follow up.
  (Only in patients who lack a SGLT-2 at inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No